CLINICAL TRIAL: NCT05876104
Title: Harassment of Pain Clinic Staff by Chronic Pain Patients
Brief Title: Harassment of Pain Clinic Staff by Patients
Status: Completed | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAne2022 Harass By Patient
Record Dates: First submitted 2023-05-11; First posted 2023-05-25 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Patient Violence
Keywords: Harassment by patients
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult chronic pain patients: Adult chronic pain patients who harass pain clinic staff
  Interventions: Behavioral: Behavioral therapy

INTERVENTIONS:
Behavioral: Behavioral therapy — Behavioral and supportive therapy

SUMMARY:
Chronic pain is associated with psychological disorders, and many patients have behavioral problems. Some patients harass pain services staff. Most healthcare staff do not report harassment by patients.

Quantitative and qualitative analysis of prospective electronic and clinic diary data. Evaluation of incidents of clinic staff harassment; caused by patients and patients' family. Analysis of causative factors, incident outcome and lessons learned.

DETAILED DESCRIPTION:
Chronic pain is associated with psychological and mental health disorders. Many patients have personality and behavioral disorders. Some patients harass their pain care providers. Most healthcare staff do not report harassment by patients.

This is a quantitative and qualitative analysis of prospective electronic and clinic diary data. It is an evaluation of incidents of pain clinic staff harassment; caused by patients and patients' family. This is an analysis of incident causative factors, incident outcome and lessons learned. The qualitative information of each incident is presented in a sensitive and careful format.

ELIGIBILITY:
Inclusion Criteria:

* adult chronic pain patients

Exclusion Criteria:

* pediatric chronic pain patients

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult chronic pain patients who are undergoing treatment in a specialist pain clinic
Sampling Method: Non-Probability Sample
Enrollment: 1102 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who harassed clinic staff | 12 months
  Percentage of patients who harassed clinic staff

CONTACTS AND LOCATIONS:
Overall Officials: Olu Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] David K, Anuj D, Nabil S. Violence toward chronic pain care providers: A national survey. Pain Med. 2015 Oct;16(10):1882-96. doi: 10.1111/pme.12794. Epub 2015 Jun 2. PMID 26037534
- [Background] Bamgbade OA, Tai-Osagbemi J, Bamgbade DO, Murphy-Akpieyi O, Fadire A, Soni NK, Mumporeze L. Clonidine is better than zopiclone for insomnia treatment in chronic pain patients. J Clin Sleep Med. 2022 Jun 1;18(6):1565-1571. doi: 10.5664/jcsm.9930. PMID 35112665
- [Background] Bamgbade OA, Onongaya V, Anomneze-Collins A, Omoniyi DA, Simmonds-Brooks P, Richards RN. Delayed surgical diagnosis and treatment of severe sickle cell arthropathy: The need to raise clinicians' awareness. J Taibah Univ Med Sci. 2021 May 31;16(5):683-688. doi: 10.1016/j.jtumed.2021.04.007. eCollection 2021 Oct. PMID 34690647
- See also: Pain Management and Sociology Implications: The Sociomedical Problem of Pain Clinic Staff Harassment Caused by Chronic Pain Patients — https://brieflands.com/articles/aapm-144263